CLINICAL TRIAL: NCT04370067
Title: Hungarian CoronaVirus Disease-19 Epidemiological Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Semmelweis University (Other); Szeged University (Other); University of Pecs (Other); University of Debrecen (Other)
Responsible Party: Sponsor
Other Study IDs: H-UNCOVER
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection
Keywords: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hungarian CoronaVirus disease-19 Epidemiological Research

DETAILED DESCRIPTION:
The planned large-scale, cross-sectional, representative population screening can show the prevalence of COVID-19 and the degree of infection and trans-infection in Hungary after more than one month of strict restriction. In addition, it can have an impact on further actions, and we can track the impact of the decisions we make by repeating the screenings.

ELIGIBILITY:
Inclusion Criteria:

* Hungarian male or female patients aged 14 and over who live in private households
* Inactivated social security number does not infer the exclusion of the study

Exclusion Criteria:

* Patients under the age of 14
* Patients living in institutional households

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hungarian male or female patients aged 14 and over who live in private households.
Sampling Method: Non-Probability Sample
Enrollment: 11200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 rate | 1 year
  The rate of the infected patients, asymptomatic carrier and healed patients

CONTACTS AND LOCATIONS:
Overall Officials: Béla Merkely, PhD,DSc, Principal Investigator — Semmelweis University Heart and Vascular Center
Locations (4):
- Hungary (4):
  - Semmelweis University - Heart and Vascular Center, Budapest
  - University of Debrecen, Debrecen
  - University of Pecs, Pécs
  - University of Szeged, Szeged

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Merkely B, Szabo AJ, Kosztin A, Berenyi E, Sebestyen A, Lengyel C, Merkely G, Karady J, Varkonyi I, Papp C, Miseta A, Betlehem J, Burian K, Csoka I, Vasarhelyi B, Ludwig E, Prinz G, Sinko J, Hanko B, Varga P, Fulop GA, Mag K, Voko Z; HUNgarian COronaVirus-19 Epidemiological Research (H-UNCOVER) investigators. Novel coronavirus epidemic in the Hungarian population, a cross-sectional nationwide survey to support the exit policy in Hungary. Geroscience. 2020 Aug;42(4):1063-1074. doi: 10.1007/s11357-020-00226-9. Epub 2020 Jul 17. PMID 32677025